CLINICAL TRIAL: NCT07197931
Title: Comparison of Circumferential Pulmonary Vein (PV) Isolation Alone Versus Additional EXtra-PulmOnaRy Vein Trigger Ablation in Persistent Atrial Fibrillation
Brief Title: EXPORT Randomized Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-1476-001
Record Dates: First submitted 2025-09-26; First posted 2025-09-30 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Additional extra-pulmonary vein trigger ablation group (Experimental): circumferential pulmonary vein isolation with additive induction, mapping, and ablation of non-pulmonary vein trigger
  Interventions: Procedure: Additional extra-pulmonary vein trigger ablation group
- Empirical pulmonary vein isolation group (Active Comparator): circumferential pulmonary vein isolation only
  Interventions: Procedure: Empirical pulmonary vein isolation group

INTERVENTIONS:
Procedure: Additional extra-pulmonary vein trigger ablation group — 1. Circumferential PVI is performed in all patients.
  2. After PVI, isoproterenol is infused starting at 5 μg/min, increased every 3-5 min to 10 and 20 μg/min (max 30 μg/min) to reach 85% of predicted heart rate for ≥10 min.
     2-1) If AF persists, internal cardioversion (5-30 J) is performed using catheters in the right atrium and coronary sinus.
     2-2) If sinus rhythm is present, a 15-beat drive train (10 mA, 2 ms) is delivered at 250 ms, shortened by 10 ms to 180 ms or until capture fails, up to three times, to induce AF or AT. Isoproterenol continues for 2 min. If arrhythmia occurs, cardioversion is repeated.
  3. After cardioversion, isoproterenol is stopped and the patient is observed for 10 min.
  4. Sustained or reproducible arrhythmias are defined as non-PV triggers.
  5. These are localized with activation mapping, P-wave analysis, and high-density mapping.
  6. Ablation is performed with the same catheter.
  7. Reassessment is done with the same protocol.
  Arms: Additional extra-pulmonary vein trigger ablation group
Procedure: Empirical pulmonary vein isolation group — 1. Circumferential pulmonary vein isolation (PVI) is performed in all patients.
  2. After PVI, a waiting period of at least 20 minutes is observed, followed by reassessment of pulmonary vein isolation before concluding the procedure.
  3. Additional linear ablation or CFAE ablation not specified in the study protocol should be avoided whenever possible.
  4. In cases where typical atrial flutter has been documented prior to the procedure or is induced during the procedure, cavo-tricuspid isthmus (CTI) ablation is performed. At the operator's discretion, CTI ablation may also be permitted even in patients without a prior history or inducibility.
  5. If atypical atrial flutter involving these pathways is induced during the procedure, additional linear ablation (e.g., roof line, posterior-inferior line, left lateral isthmus, or anterior line) may be performed.
  Arms: Empirical pulmonary vein isolation group

SUMMARY:
Pulmonary Vein Isolation (PVI)-Only Group

1. Pulmonary vein isolation (PVI) will be performed, and the procedure will be terminated without the administration of isoproterenol following the standard waiting period.
2. In cases where spontaneous triggers are observed following PVI, mapping and ablation of the identified triggers are permitted.
3. Post-procedural rhythm monitoring and follow-up will be conducted in accordance with the predefined study protocol.

Additional Non-Pulmonary Vein (Non-PV) Trigger Ablation Group

Isoproterenol will be administered starting at 5 μg/min, with stepwise increases to 10 μg/min and 20 μg/min at 3-5 minute intervals, as tolerated, aiming to achieve 85% of the maximum predicted heart rate, with a maximum dose of 30 μg/min.The total infusion duration will be at least 10 minutes.

* If systolic blood pressure (SBP) decreases by ≥20 mmHg from the baseline (prior to infusion), the isoproterenol infusion will be discontinued.
* If hypotension is anticipated or occurs during isoproterenol infusion, phenylephrine infusion may be administered to maintain SBP between 120-140 mmHg.
* For patients with a history of coronary artery disease, heart failure, or valvular heart disease, the maximum isoproterenol infusion rate may be limited to ≤10 μg/min at the discretion of the operator.

DETAILED DESCRIPTION:
"A. Essential Standard Pre-Procedural Examinations for Catheter Ablation

* Transthoracic Echocardiography (TTE): Performed in all patients to evaluate the presence of structural heart disease, left atrial size, and left ventricular function. Findings guide the selection of antiarrhythmic medications and assist in determining procedural indications.
* Transesophageal or Intracardiac Echocardiography: Conducted in all patients prior to the procedure to detect thrombi within the left atrial appendage, thereby minimizing the risk of post-procedural cerebrovascular events.
* Three-Dimensional Cardiac CT Imaging (substitutable with Cardiac Magnetic Resonance Imaging if clinically indicated): Performed in all patients before the procedure to generate a three-dimensional anatomical model of the left atrium by integrating voltage mapping and contour data from CT images. This approach enhances procedural accuracy and reduces the incidence of procedure-related complications.
* The most recent test results prior to the procedure should be utilized preferentially; in the absence of recent data, prior examination results may be used as substitutes.

B. Administration of Medications Before and After Catheter Ablation

* Anticoagulant therapy will be administered for a period of one month prior to and for a minimum of two months following the catheter ablation procedure, in order to reduce the risk of thromboembolic events, including stroke. Should the risk of stroke remain elevated due to atrial fibrillation recurrence or other clinical considerations, continuation of anticoagulation therapy may be determined at the discretion of the treating physician.
* In cases where recurrence of atrial fibrillation is suspected, or if there is a clinically assessed high likelihood of recurrence, antiarrhythmic medications may be prescribed based on the clinical judgment of the physician.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥19 years with persistent atrial fibrillation scheduled for catheter ablation.
* Refractory to or intolerant of at least one Class I or III antiarrhythmic drug.
* Undergoing first-time catheter ablation for atrial fibrillation.

Exclusion Criteria:

* Acute coronary syndrome within the past 3 months.
* Severe unrevascularized coronary artery disease: ≥70% stenosis in at least one major epicardial vessel with a diameter ≥2 mm.
* History of stroke or transient ischemic attack (TIA) within the past 3 months.
* Uncontrolled severe hypertension (systolic blood pressure ≥180 mmHg or diastolic blood pressure ≥120 mmHg).
* Severe untreated aortic valve stenosis.
* Symptomatic moderate-to-severe valvular heart disease.
* Aortic dissection.
* Heart failure with reduced ejection fraction (LVEF <40%).
* Severe pulmonary hypertension (resting RVSP >60 mmHg).
* Left atrial anteroposterior diameter >60 mm.
* Presence of cyanotic congenital heart disease.
* Obstructive hypertrophic cardiomyopathy (resting or provoked LVOT pressure gradient ≥30 mmHg).
* History of prior maze surgery or catheter ablation for atrial fibrillation.
* Active internal bleeding.
* Contraindications to anticoagulation therapy or rhythm control treatment.
* Presence of severe comorbid conditions or life expectancy <1 year.
* Drug or alcohol abuse.
* Pregnancy.
* Any other condition that, in the investigator's judgment, makes the patient unsuitable for study participation.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 406 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2029-08-31 (Estimated); Study Completion 2030-08-31 (Estimated)

PRIMARY OUTCOMES:
Recurrence of atrial arrhythmia | within 24 months after enrollement
  any documented atrial arrhythmia lasting ≥30 seconds after a 3-month blanking period following ablation with or without the use of antiarrhythmic drug use

SECONDARY OUTCOMES:
Recurrence of atrial arrhythmia or use of antiarrhythmic drug | within 24 months after enrollement
  any documented atrial arrhythmia lasting ≥30 seconds after a 3-month blanking period following ablation or the use of antiarrhythmic drug use
Recurrence of atrial fibrillation | within 24 months after enrollement
  any documented atrial fibrillation lasting ≥30 seconds after a 3-month blanking period following ablation with or without the use of antiarrhythmic drug use
Recurrence of atrial tachycardia/flutter | within 24 months after enrollement
  any documented atrial tachycardia/flutter lasting ≥30 seconds after a 3-month blanking period following ablation with or without the use of antiarrhythmic drug use
Cardioversion rate | within 24 months after enrollement
  any cardioversion performed following ablation
Complication rate | within 24 months after enrollement
  any complication related to ablation

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Cardiovascular Hospital, Yonsei University Health System, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided